CLINICAL TRIAL: NCT00235066
Title: A Multicenter, Nonrandomized, Historical Controlled Study In Patients With De Novo Coronary Artery Lesions In Small VessELs Treated With The CYPHER™ STEnt
Brief Title: The CYPHER™ Stent Study in Patients With Small de Novo Coronary Artery Lesions.
Acronym: SVELTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll, MD, Cordis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC02-04
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Cypher Sirolimus-Eluting Stent
  Interventions: Device: PCI

INTERVENTIONS:
Device: PCI — PCI with Cypher Sirolimus-Eluting Stent
  Other Names: drug-eluting stent

SUMMARY:
The main objective of this study is to assess the effectiveness of the CYPHER™ (sirolimus-eluting) stent in reducing in-lesion late lumen loss in de novo native coronary artery lesions in small vessels (2.25 - 2.75 mm) as compared to the small vessel tercile of the uncoated Bx VELOCITYTM Stent patients from the SIRIUS Trial, using a stenting technique that minimizes balloon trauma to the vessel and assures full coverage of the lesion with the stent.

DETAILED DESCRIPTION:
This is an international, multicenter (up to 10 sites), nonrandomized, historically controlled study in patients with De Novo coronary artery lesions in small vessels treated with the CYPHER™ (sirolimus-eluting) stent as compared to the small vessel tercile uncoated Bx VELOCITYTM Stent patients from the SIRIUS Trial. A total of up to 100 patients will be enrolled in this study.

Patients with de novo native coronary artery lesions >=15mm and <=30mm in length and >=2.25 mm to <=2.75 mm in diameter by visual estimation will be treated with the CYPHER™ (sirolimus-eluting) stent. Patients will be followed at 30 days, 6, 8, 9 months and at 1, 2 and 3 years post-procedure, with a repeat angiography at 8 months. In all patients Intravascular Ultrasound (IVUS) will be performed before (only in case of crossing success) and after the initial procedure. An IVUS control will also be done at 8 months follow up to assess neo-intimal growth and remodeling.

This is a single lesion treatment study. Patients may have other lesions treated before the treatment of the intended lesion in the small vessel (a non-target lesion may not be located in the target vessel!). Post-procedural treatment of another lesion is only allowed after the 30-day follow-up contact has been completed or in case this is clinically needed.

It is anticipated that the total length of the study will be 39 months: 3 months to complete patient enrollment and 3 years for follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS 1, 2, 3, 4) OR unstable angina pectoris (Braunwald Classification B&C 1-2) OR patients with documented silent ischemia;
2. Single treatment of de novo lesion in a small vessel (2.25 - 2.75 mm) in a major coronary artery in patients with single or multivessel disease. Patients with multiple lesions can be included if the other lesions are successfully treated prior to the treatment of the intended lesion in the small vessel.
3. Target vessel diameter >=2.25 and <=2.75mm (by visual estimation);
4. Target lesion length >=15 and <=30 mm.

Exclusion Criteria:

1. Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK >2 times normal within the preceding 24 hours or the CK and CK-MB remains above normal at the time of the treatment;
2. Has unstable angina classified as Braunwald A (1, 2, 3) or B & C 3;
3. Unprotected left main coronary disease with >=50% stenosis;
4. Significant (>50%) stenosis proximal or distal to the target lesion that might require revascularization or impede inflow or runoff;
5. Have an ostial target lesion;
6. Lesion < 2.25 or > 2.75 mm in diameter;
7. Totally occluded vessel (TIMI 0 level);
8. Documented left ventricular ejection fraction £30%;
9. Intention to treat the target lesion by direct stenting procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-11; Primary Completion 2003-11 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
In-lesion late lumen loss | 8-moths post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Meier, MD, Principal Investigator — University of Bern
Locations (1):
- University Hospital, Swiss Cardiovascular CenterBern, Bern, Switzerland

REFERENCES:
- [Result] Meier B, Sousa E, Guagliumi G, Van den Branden F, Grenadier E, Windecker S, te Riele H, Voudris V, Eltchaninoff H, Lindvall B, Snead D, Talen A; SVELTE Study Group. Sirolimus-eluting coronary stents in small vessels. Am Heart J. 2006 May;151(5):1019.e1-7. doi: 10.1016/j.ahj.2006.02.025. PMID 16644326